CLINICAL TRIAL: NCT02575989
Title: Prevention of HYPOthermia Before Admission in TRAUMa Patients - Hypotraum 2 Study
Brief Title: Prevention of HYPOthermia in TRAUMa Patients
Acronym: HYPOTRAUM 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 131204; 2014-A00564-43 (Other: IDRCB)
Record Dates: First submitted 2015-09-15; First posted 2015-10-15 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Trauma Patients
Keywords: Trauma; Prehospital; Hypothermia
MeSH Terms: conditions — Wounds and Injuries; Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: control group (Active Comparator): Classic - current management of trauma patients by French medical teams
  Interventions: Other: 1: control group
- 2: interventional group (Experimental): Intervention Name : monitoring, treatment, control and prevention of hypothermia
  * Continuous monitoring of body temperature
  * Ambulance warming (target : 30°C)
  * Patient warming with dedicated blanket
  * Infusion fluid warming (and temperature control)
  Interventions: Other: 2: interventional group

INTERVENTIONS:
Other: 1: control group — Classic - current management of trauma patients by French medical teams
  Arms: 1: control group
Other: 2: interventional group — Intervention Name : monitoring, treatment, control and prevention of hypothermia
  * Continuous monitoring of body temperature
  * Ambulance warming (target : 30°C)
  * Patient warming with dedicated blanket
  * Infusion fluid warming (and temperature control)
  Arms: 2: interventional group

SUMMARY:
The purpose of this study is to demonstrate that the specific management will increase the number of alive trauma patient arriving with a temperature > 35°C.

DETAILED DESCRIPTION:
Trauma patients are often hypothermic (temperature < 35 °C) upon arrival at the hospital. Hypothermia is with hypotension and hypoxia, perfectly known to be directly responsible for complications.

Hypothermia is responsible, with acidosis and coagulopathy, of the " lethal triad" of trauma.

Thus, it is clearly established that hypothermia is directly associated with poor prognostic in trauma patients. In a recent study, mortality rate reached 100% for trauma patients arriving at the hospital with a body temperature below 32°C.

The weather, the severity of the trauma and medical (or paramedical) interventions are responsible for the onset of this hypothermia.

Then, continuous monitoring of the patient's temperature, active protection against hypothermia with a metal blanket, the warming (and measure the temperature of) infusion fluids, the warming (and measure the temperature of) the ambulance should improve patient's outcome. As hypothermia is associated with mortality of trauma patients, the control must lead to reduce mortality.

Randomization Due to the use of a global management strategy with combination of several specific interventions and the need for special equipment (heating devices infusion fluids), randomization will be done by investigator center: interventional center (combining the different interventions) and standard management (without modification, except measurements of the patient's and air temperature at inclusion and on arrival at a receiving center.

In this context, it is also crucial that the weather conditions, the characteristics of trauma and patients were similar in both groups. Also, 12 investigation centers will be classified based on annual local average temperatures.

Main collected data Demographics and morphological traits (age, sex, body weight, and height of the victim), the nature and circumstances of the accident (date, time, place), the victim's presentation on mobile intensive care unit (MICU) arrival (trapped or not, seated or lying down, on the ground, unclothed, wet, or covered by a blanket, environmental conditions, clinical factors, and care provided.

Environmental conditions included air (indoors or outdoors) temperature, and rain at the site of the accident as well as mobile intensive care unit temperature.

Clinical factors included: the site and nature of the lesions (fracture, wound, contusion), heart rate, the Revised Trauma Score (RTS) (Glasgow Coma Score (GCS) + systolic blood pressure + respiratory rate), oxygen saturation or oxygen delivery, and tympanic temperature.

Whenever applicable: vascular filling (infusion fluid temperature and volumes), catecholamine and morphine administration, any other drugs (with doses), orotracheal intubation.

Times from the accident to MICU arrival and from MICU arrival to hospital admission.

Statistical analysis Primary endpoint: rate of patients arriving at the hospital with a temperature <35°C. These data will be analyzed by model of multi-level logistic regression to again consider the cluster design of the study. A secondary analysis will enter the model known a priori factors that may affect hypothermia. The parameters corresponding to the secondary objectives will be entered in a model of logistic regression multivariate thereby specifically test their effect on the criteria studied.

Secondary endpoints: Binary secondary endpoints will be analyzed by model of multi-level logistic regression. Quantitative secondary endpoints will be analyzed by mixed model ANCOVA introducing randomness in the center. The variables may be processed before analysis for non-Gaussian distribution. In case of failure of the normalizing transformation, exact procedure may be used.

Number of patients to include The calculation of the sample size was based on our previous study.* The incidence of hypothermia on arrival at the hospital was 14%. By selecting high-risk patients, the investigators expect an incidence of about 20%. The objective is to achieve a reduction of one third of hypothermia (i.e. from 20 to 13 %). Using a two-tailed test at α risk of 0.05 and 1 - beta 0.8, the calculation of required number of patients is 440 per group. Assuming a moderate inflation factor of about 1.35 related to the cluster randomization (our experience shows that intra-cluster correlation coefficients are low) the total number of patients per group will be 600 patients.

A total of N = 1,200 patients for the study.

ELIGIBILITY:
Inclusion criteria :

* Patient with trauma (> 18 years)
* Pre-hospital management by MICU
* Scheduled transfer to a receiving center by a MICU
* And at least one of the following criteria :

  * Ambient temperature on the field < 18°C
  * Body temperature <35°C on MICU arrival
  * A Glasgow score < 15 on MICU arrival
  * Systolic blood pressure < 100 mm Hg on MICU arrival

Exclusion criteria :

- Body temperature <31°C or >38°C

* Cardiac arrest before MICU arrival
* Bilateral ear bleeding preventing continuous monitoring of tympanic temperature

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1086 (Actual)
Dates: Start 2016-01-17 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Number of trauma patients arriving alive with a temperature > 35°C (at receiving hospital) | Day0

SECONDARY OUTCOMES:
Survival at hospital discharge | up to 3 months
Length of stay at hospital (days) | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric LAPOSTOLLE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- SAMU 93, AP-HP, Urgences - SAMU 93, Unité Recherche-Enseignement-Qualité, Hôpital Avicenne, Bobigny, France

REFERENCES:
- [Background] Lapostolle F, Sebbah JL, Couvreur J, Koch FX, Savary D, Tazarourte K, Egman G, Mzabi L, Galinski M, Adnet F. Risk factors for onset of hypothermia in trauma victims: the HypoTraum study. Crit Care. 2012 Jul 31;16(4):R142. doi: 10.1186/cc11449. PMID 22849694